CLINICAL TRIAL: NCT07077980
Title: Discovery of HPV T Cell Epitopes and Development of Multi-epitope Vaccines
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: YingZhou 2025-3
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on the trend that the incidence and mortality of cervical carcinoma among female cancers worldwide are increasing year by year, the investigators aim to develop a multi-epitope therapeutic vaccine capable of simultaneously activating humoral and cellular immune responses, which is achieved by fusing multiple T-cell epitope immunostimulatory proteins. To obtain information on functional T-cell epitopes to be included in the vaccine, the investigators conducted research starting from clinical cases. By collecting peripheral blood and cancerous tissues from clinical patients, the investigators isolated reactive T-cells and screened for information on T-cell epitopes of HPV antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged between 18 and 65 who can receive standard treatment, including those who only undergo surgery or those who receive radiotherapy and chemotherapy after surgery.
2. Cervical carcinoma caused by HPV16 or HPV18 infection.
3. The pathological stage is from IB1 to IV, and informed consent is obtained.
4. If the tumor tissue of patients with stage IB1 is not obvious, samples can be taken or not taken without affecting subsequent pathological examinations.

Exclusion Criteria:

1. Patients with other malignancies
2. Patients with any uncontrolled systemic disease, including active infection, uncontrolled hypertension, diabetes mellitus, unstable angina and congestive heart failure, myocardial infarction (1 year) before starting treatment, severe arrhythmia requiring medical treatment, coagulation abnormalities, liver or kidney or metabolic disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients diagnosed with HPV16 or HPV18 infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
The activity of T cell | one month
  The T cell activity exceeds 95%.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No